CLINICAL TRIAL: NCT02147496
Title: The Effect of Fluid Dairy Products Consumed Before and Within a Pizza Meal on Glycemic Regulation, Food Intake and Satiety in Normal Weight and Overweight/Obese Children
Brief Title: Fluid Dairy Products Consumed Before and Within a Pizza Meal on Glycemic Response, Food Intake and Satiety in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Dairy Farmers of Canada (Other); The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: DFC kids 25804; DFC Kids Milk Study 491336
Record Dates: First submitted 2013-12-09; First posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Prevention; Obesity Prevention
Keywords: Food intake; Appetite; Blood glucose; Insulin; Dairy; Milk
MeSH Terms: conditions — Insulin Resistance | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 2% M.F. Milk (Experimental): Dietary treatment: 2% m.f. milk
  Interventions: Other: Dietary Intervention
- 1% M.F. Chocolate Milk (Experimental): Dietary treatment: 1% m.f. chocolate milk
  Interventions: Other: Dietary Intervention
- 1.5% M.F. Drinkable Yogurt (Experimental): Dietary treatment: 1.5% m.f. drinkable yogurt
  Interventions: Other: Dietary Intervention
- Tropical Punch (Experimental): Dietary treatment: fruit-flavoured beverage
  Interventions: Other: Dietary Intervention
- Water (Experimental): Dietary treatment: calorie-free control
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention

SUMMARY:
The purpose of this study is to examine the effects of fluid dairy products on blood glucose and insulin, satiety and energy intake in normal weight and overweight/obese children in the age range of 9-14 y. Experiment 1: The specific objective is to examine the effects of isocaloric and isovolumetric amounts of 2% M.F. milk, 1% M.F. chocolate milk, 1.5% M.F. yogurt drink, tropical punch and water consumed before and within a pizza meal 60 min later on appetite and food intake. Experiment 2 will compare the effects of 2% M.F. milk and tropical punch consumed before and with a pizza meal 60 min later on food intake, blood glucose, and appetite hormone response.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Born at term

Exclusion Criteria:

* Diabetes
* Medications
* Lactose-intolerance or allergies to milk
* Breakfast skippers and those on an energy restricted diet

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Food intake | 60 minute
  The amount of food (grams) and energy (kcal) consumed ad libidum with the test meal.

SECONDARY OUTCOMES:
Blood glucose | 0, 30, 60, 85, 115, and 145 minute
Appetite hormones | 0, 30, 60, 85, 115, and 145 minute
  Insulin, total ghrelin, glucagon-like peptide-1, and peptide YY

OTHER OUTCOMES:
Subjective Appetite | 0, 10, 20, 30, 60, 85, 95, 105, 115, and 145 minuites

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Anderson, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada